CLINICAL TRIAL: NCT03595280
Title: Optimizing Risk Messages for Waterpipe Tobacco Cessation in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Darren Mays, Assistant Professor of Oncology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1378; R01CA217861 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-23 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hookah Smoking
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Intervention Model Description: This is a randomized trial with 3 groups: 1) Control group that receives no study messages; 2) Untailored message group that receives general messages about the risks of hookah tobacco; 3) Tailored message group that receives messages about the risks of hookah tobacco that are personalized to their hookah tobacco use behavior and beliefs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in the control group receive no study messages
- Untailored Messages (Experimental): Participants in the untailored message group receive mobile multimedia service messages conveying the risks of hookah tobacco on their mobile phones.
  Interventions: Behavioral: Hookah tobacco risk messages
- Tailored Messages (Experimental): Participants in the tailored message group receive mobile multimedia service messages conveying the risks of hookah tobacco on their mobile phones that are personalized to their hookah tobacco use behavior and beliefs.
  Interventions: Behavioral: Hookah tobacco risk messages

INTERVENTIONS:
Behavioral: Hookah tobacco risk messages — Mobile multimedia messages consisting of text and imagery conveying the risks of hookah tobacco use.
  Arms: Tailored Messages; Untailored Messages

SUMMARY:
The objective of this study is to examine whether messages conveying the harms and addictiveness of waterpipe (i.e., hookah) tobacco delivered by mobile phone multimedia messaging (MMS) are effective for promoting hookah tobacco cessation among young adults ages 18 to 30 years.

DETAILED DESCRIPTION:
The purpose of this study is to test the effects of messages communicating the risks (i.e., health harms, addictiveness) of hookah tobacco delivered via mobile multimedia messaging for promoting hookah tobacco cessation. The study will also compare two messaging approaches, a standard untailored approach where all participants receive the same message content, and a tailored messaging approach where message content is personalized to baseline measures of hookah tobacco use behavior and beliefs and interactively to exchanges that occur via mobile messaging sent and received during the exposure period. The study includes young adults ages 18 to 30 who are current hookah tobacco smokers. Eligible participants are young adults ages 18 to 30 years who have smoked hookah tobacco at least once in the past month, smoke hookah tobacco on at least a monthly basis, and have access to the internet and a personal mobile phone to complete study procedures. Study participants will complete a baseline survey online, and all participants will receive standard information about the risks of hookah tobacco. Then participants will be randomly assigned to one of three groups: control group, untailored message group, tailored message group. Participants in the untailored and tailored message group will receive messages sent to their mobile phones communicating the risks of hookah tobacco for a 6 week period. All participants will complete follow-up surveys online 6 weeks after baseline, 3 months later, and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30
* Smoked hookah tobacco within the last 30 days and smokes hookah tobacco on at least a monthly basis
* Has access the internet to complete study procedures
* Has personal mobile phone to complete study procedures

Exclusion Criteria:

* Age less than 18 or greater than 30
* Has not smoked hookah tobacco in the last 30 days or does not smoke hookah tobacco on at least a monthly basis
* Does not have access to the internet to complete study procedures
* Does not have a personal mobile phone to complete study procedures

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 349 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mays, PhD, MPH, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
We will consider requests to share de-identified individual participant data by request and according to the investigator's study protocol and institutional data sharing policy.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Untailored Messages | Tailored Messages
Started | 119 | 117 | 113
Completed | 113 | 108 | 98
Not Completed | 6 | 9 | 15
Not completed — Lost to Follow-up | 6 | 9 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Untailored Messages | Tailored Messages | Total
Number analyzed (Participants) | 119 | 117 | 113 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (3.4) | 23.7 (3.5) | 24.6 (3.5) | 24.0 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 57 | 59 | 187
  Male | 48 | 60 | 54 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 11 | 40
  Not Hispanic or Latino | 104 | 103 | 101 | 308
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Asian | 8 | 14 | 9 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 1 | 5
  Black or African American | 27 | 26 | 27 | 80
  White | 51 | 43 | 53 | 147
  More than one race | 30 | 31 | 21 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Less Than College Education | 16 | 24 | 16 | 56
  Some College or Higher | 103 | 93 | 97 | 293

OUTCOME MEASURES:

1. Primary Outcome: Perceived Harm
Description: Perceived harm of hookah tobacco is measured using valid self-report item assessing perceptions of how likely harms are to occur from hookah tobacco use (response range 1 no chance to 7 certain to happen). Greater perceived likelihood of harm is considered a better outcome. The assessment is administered immediately post intervention, 3-month follow-up, and 6-month follow-up, 6 month follow-up data reported.
Time Frame: 6-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
score on a scale | 4.1 [3.9 to 4.4] | 4.2 [4.0 to 4.5] | 4.5 [4.2 to 4.8]

2. Primary Outcome: Perceived Addictiveness
Description: Perceived addictiveness of hookah tobacco is measured using valid self-report item assessing perceptions of how likely one is to become addicted to hookah tobacco (1 = no chance, 7 = certain to happen). Greater perceived likelihood of addictiveness is considered a better outcome. The assessment is administered immediately post-intervention, 3-month follow-up, and 6 month follow-up, 6-month follow-up data reported.
Time Frame: 6-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
score on a scale | 3.9 [3.5 to 4.2] | 3.9 [3.6 to 4.3] | 4.0 [3.7 to 4.3]

3. Primary Outcome: Worry About Harm
Description: Worry about the harms of hookah tobacco is measured using a valid self-report item assessing how much participants worry about the risks of hookah tobacco (1 = Not at all, 7 = Very much). Greater worry about harm is considered a better outcome. The assessment is administered immediately post-intervention, 3-month follow-up, and 6 month follow-up, 6-month follow-up reported.
Time Frame: 6-months
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
score on a scale | 4.6 [4.3 to 5.0] | 4.1 [3.8 to 4.5] | 4.6 [4.3 to 5.0]

4. Primary Outcome: Worry About Addictiveness
Description: Worry about the addictiveness of hookah tobacco is measured using a valid self-report item assessing how much participants worry about becoming addicted to hookah tobacco (1 = Not at all, 7 = very much). Greater perceived addictiveness is considered a better outcome. The assessment is administered immediately post-intervention, 3 month follow-up, and 6 month-follow-up, 6 month follow-up reported.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
score on a scale | 3.6 [3.2 to 3.9] | 3.7 [3.3 to 4.1] | 3.9 [3.5 to 4.3]

5. Primary Outcome: Motivation to Quit
Description: Motivation to quit is measured using a valid self-report item assessing how much participants want to quit smoking hookah tobacco right now (1 = Not at all, 7 = Very). Greater motivation to quit is considered a better outcome. The assessment is administered immediately post-intervention, 3 month follow-up, and 6 month follow-up, 6-month follow-up reported.
Time Frame: 6-months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
units on a scale | 4.0 [3.5 to 4.4] | 4.0 [3.5 to 4.4] | 3.5 [3.0 to 4.1]

6. Primary Outcome: Hookah Tobacco Use Frequency
Description: Hookah tobacco use frequency is measured using a valid self-report item assessing how often participants have smoked hookah tobacco in the past 30 days. The item measures the number of days in the past month participants have smoked hookah tobacco. Less frequent hookah tobacco use is considered a better outcome. The assessment is administered immediately post-intervention, 3 month follow-up, and 6 month follow-up, 6-month follow-up reported.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: days in the past month
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
days in the past month | 4.3 [3.0 to 5.6] | 4.0 [2.6 to 5.2] | 3.5 [2.0 to 5.0]

7. Primary Outcome: Percent of Participants Who Quit Smoking Hookah Tobacco
Description: Hookah tobacco cessation is measured using a single valid self-report item assessing if participants have stopped smoking hookah tobacco completely. The item asks if participants have completely stopped smoking hookah tobacco based on a yes/no response. Quitting hookah tobacco use (i.e., responses of "yes") is considered a better outcome. The assessment is administered immediately post intervention, 3 month follow-up, and 6 month follow-up, 6-month follow-up data reported.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Control | Untailored Messages | Tailored Messages
Number analyzed (Participants) | 113 | 108 | 98
percentage of participants | 29.20 | 37.96 | 48.98

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control | Untailored Messages | Tailored Messages
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/108 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/108 | 0/98
Other Adverse Events (participants affected / at risk) | 0/113 | 0/108 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03595280/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03595280/SAP_001.pdf